CLINICAL TRIAL: NCT07250711
Title: Effect of Anal Lift Exercise on Rehabilitation After Anal Fistula Surgery: a Single-center, Prospective, Open-label, Randomized Clinical Trial
Brief Title: Effect of Anal Lift Exercise on Rehabilitation After Anal Fistula Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Putian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PutianU-007
Record Dates: First submitted 2025-09-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Kegel Exercises
Keywords: anal fistula; Kegel Exercise
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation group (No Intervention): Explain the relevant postoperative precautions and instructions to the patients, and the observation group is allowed to perform random movements.
- Control group (Experimental): Explain the relevant postoperative precautions and instructions to the patients, and have the control group perform pelvic floor contraction exercises.
  Interventions: Procedure: Kegel exercises

INTERVENTIONS:
Procedure: Kegel exercises — The patient carried out pelvic floor elevation exercises after the surgery, aiming to accelerate the recovery process and alleviate the pain.
  Arms: Control group

SUMMARY:
Anorectal fistula refers to a granulomatous duct located around the rectum and anus. It is mostly caused by infection of the soft tissues surrounding the rectum and anus, and often presents with symptoms such as swelling, pain, and itching around the anus. This causes inconvenience to the patient's daily life. The ideal surgical treatment for anorectal fistula should eliminate sepsis and promote the healing of the duct, while preserving the sphincter and the defecation mechanism. Abbas mentioned the predictive factors for postoperative results of anorectal fistula. Some sinus tracts are relatively deep, the surgical scope is relatively large, the destruction of the rectal ring, which causes a significant feeling of anal distension, will affect the defecation function. After the operation, effective intervention measures should be taken to promote the patient's recovery. Kegel exercise, also known as pelvic floor exercise, is a regular upward lifting and contraction of the anus. It can promote peripheral blood circulation, relieve pain, improve the function of the anal sphincter, and also enhance the strength around the anus to prevent the occurrence of anal incontinence. It is mainly used for the treatment and improvement of anal diseases. When patients perform pelvic floor exercises, they should also pay attention to a light diet and avoid using spicy and irritating foods to avoid affecting the effect of the pelvic floor exercise. Combined with the new pain management concept of this department, for postoperative patients with anorectal fistula, pelvic floor exercise intervention is carried out for constipation and anal heaviness, and the efficacy is observed.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 55 years old
* Patients diagnosed with anal fistula through digital rectal examination and anoscopy
* Receive operation

Exclusion Criteria:

* The patient has a mental disorder.
* Patients with hemorrhoids
* Anal fistula combined with perianal abscess
* Patients who are unable to cooperate with follow-up visits

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Record pain score | Day 1，2，3，4，5
  Assessment timepoints: At postoperative days 1, 2, 3, 4, 5.
Record the bleeding score. | Day 1，2，3，4，5
  Assessment timepoints: At postoperative days 1, 2, 3, 4, 5.
Record the score of anal distension and fullness. | Day 1, 2, 3, 4, 5
  Assessment timepoints: At postoperative days 1, 2, 3, 4, 5.

SECONDARY OUTCOMES:
Compare the defecation situation of the patients. | Within 30 days postoperatively
  Patients with anal fistula should start doing pelvic floor exercises and controlling their diet from the day of surgery until the fifth day. Observe the defecation situation.
Length of hospital stay | Daily from Day 1 (max 60 days post-op)
  Record the length of the patient's hospital stay and make a comparison